CLINICAL TRIAL: NCT07208786
Title: Randomized Clinical Trial on Pre-emptive Endoscopic Vacuum Therapy Versus Conventional Management for the Prevention of Anastomotic Leakage After Colorectal Cancer Surgery
Brief Title: Pre-emptive Endoscopic Vacuum Therapy Reduces the Incidence of Anastomotic Leakage After Colorectal Cancer Surgery: a Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025166
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Colorectal Surgery; Complications; Anastomotic Leakage; Endoscopic Vacuum Therapy
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-emptive Endoscopic Vacuum Therapy (Experimental): After the anastomosis is completed and confirmed by endoscopy to be intact and free of bleeding, immediately perform Pre-emptive Endoscopic Vacuum Therapy(PEVT).
  Interventions: Device: PEVT
- No Pre-emptive Endoscopic Vacuum Therapy (No Intervention): After the anastomosis, only routine colonoscopy was performed without PEVT device, and other steps were consistent with the PEVT group.

INTERVENTIONS:
Device: PEVT — PEVT Procedures
  After the anastomosis is completed and endoscopy confirms that the anastomotic site is intact and without bleeding, the following procedures are carried out immediately (usually within 30 minutes after the completion of the anastomosis):
  1. EVT device selection: Use an open-pore polyurethane sponge (OPPS) connected to a 16Fr nasogastric tube, with the sponge cut to a size of 2 cm × 3 cm.
  2. Placement method: Insert the sponge through the anus to the anastomotic site in the intestinal lumen, set the negative pressure to low intensity (-50 to -100 mmHg), and connect to an external negative pressure suction device for continuous suction.
  Arms: Pre-emptive Endoscopic Vacuum Therapy

SUMMARY:
Evaluate the safety and efficacy of postoperative Pre-emptive EVT (PEVT) in reducing the incidence of anastomotic leaks within 30 days after surgery in patients with colorectal cancer. Compare the differences between the PEVT group and the control group in terms of operation time, length of hospital stay, and total medical costs. Analyze the incidence of other postoperative complications in the two groups, such as wound infection, abdominal abscess, and intestinal obstruction. Assess the impact of PEVT on postoperative recovery indicators, including time to first flatus, time to first defecation, and time to ambulation. Observe the occurrence of PEVT-related adverse events, such as device displacement, bleeding, and infection.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed with colorectal cancer, planned for radical surgery (right hemicolectomy, left hemicolectomy, or anterior resection of the rectum, etc.).
2. Age 18-85 years, American Society of Anesthesiologists (ASA) classification I-III.
3. Anastomosis to be performed in a single stage (meeting anastomotic criteria).
4. Patient or legal guardian is able to understand and sign the informed consent form and comply with follow-up.

Exclusion Criteria:

1. Preexisting anastomotic leakage or severe intra-abdominal infection before surgery.
2. Complicated by severe cardiovascular or cerebrovascular diseases (e.g., acute myocardial infarction, acute phase of cerebral infarction).
3. Severe liver or kidney dysfunction (liver function Child-Pugh class C, creatinine clearance <30 ml/min).
4. Coagulation disorders (platelets <50×10⁹/L, INR >1.5) or receiving anticoagulant therapy that cannot be adjusted.
5. History of abdominal radiotherapy or multiple abdominal surgeries leading to severe intra-abdominal adhesions.
6. Complicated by other malignant tumors and currently undergoing radiotherapy or chemotherapy.
7. Psychiatric illness or cognitive impairment preventing compliance with the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Anastomotic Leak within 30 days | 30 days
  Count the number of participants who develop anastomotic leak within 30 days after colorectal cancer surgery.

SECONDARY OUTCOMES:
Number of Participants with Postoperative Complications within 30 days | 30 days
  Count the number of participants who develop postoperative bleeding, anastomotic stenosis, and intra-abdominal infection within 30 days after colorectal cancer surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchong Central Hospital, Nanchong, Sichuan, China